CLINICAL TRIAL: NCT01321801
Title: Preoperative Use of Pregabalin and Analgesia Levels After Laparoscopic Cholecystectomy
Brief Title: Pregabalin and Analgesia After Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Larissa University Hospital (Other)
Responsible Party: Principal Investigator, Chamaidi Sarakatsianou, RN,MSc, Larissa University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UHL25872/ 08/17/09
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Pain Postoperative
Keywords: Pregabalin; Laparoscopic cholecystectomy; Postoperative pain; Opioid consumption
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pregabalin (Active Comparator): Preoperative administration of pregabalin 600mg to patients undergo laparoscopic cholecystectomy.Patients receive oral Pregabalin 300 mg the night before the surgery, and another one dose of 300 mg 1 hour prior to surgery
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator): Preoperative administration of placebo to patients undergo laparoscopic cholecystectomy.Patients receive oral Placebo the night before the surgery, and another one dose 1 hour prior to surgery.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Pregabalin — Preoperative administration of pregabalin 600mg
  Other Names: Lyrica
  Arms: Pregabalin
Drug: placebo — Preoperative administration of a matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate how effective is the preoperative administration of pregabalin 600mg, to attenuate postoperative pain and opioids consumption after laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Acute pain frequently occurs during the postoperative period.Not treated acute postoperative pain may predict the development of chronic pain.Recently, the analgesic effect of pregabalin, as a part of a multimodal analgesia, has been evaluated in many studies. They have shown that pregabalin may have a role in the post operative pain management, as an adjunct. Pregabalin is an anticonvulsant and anxiolytic drug, which have a more favorable pharmacokinetic profile from its predecessor gabapentin.

Acute postoperative pain after laparoscopic cholecystectomy is complex in nature. Postoperative pain is the main complaint and the primary reason for delay discharge after laparoscopic cholecystectomy.The study includes patients undergoing laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II

Exclusion Criteria:

* Renal or hepatic insufficiency
* Alcohol or drugs abuse
* History of chronic pain or daily intake of analgesics
* Uncontrolled medical disease (hypertension, diabetes) and cardiovascular problems. Psychiatric disorders
* Inability of patients to use PCA pump
* History of intake of non-steroidal anti-inflammatory drugs the last 24 hours before surgery,use of drainage after the surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-11; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | Every 8 hours
  VAS = visual analoque scale 0-10 mm (0=no pain to 10= worst imaginable pain).Measured on the arrival of the patient to the recovery room(0 hrs), one hour later, and then every eight hours until the completion of 24 hours after operation.

SECONDARY OUTCOMES:
Side- effects | 0,1, 8, 16 & 24 hours
  To determine the occurrence of side effects such as postoperative nausea,vomiting, itching, headache, dizziness, blurred vision, lack of concentration, shoulder pain, sedation, and respiratory depression.
Postoperative opioid consumption | 0,1, 8, 16 & 24 hour
  The total dose of morphine was calculated as mg and included opioids administered by PCA pump.On arrival in the PACU patients received morphine via PCA pump.Postoperative morphine requirements were assessed on the arrival of the patient to the recovery room (0 hrs), one hour later and then every eight hours, until the completion of 24 hours after operation.

CONTACTS AND LOCATIONS:
Overall Officials: Chamaidi Sarakatsianou, RN, MSc, Principal Investigator — University Hospital of Larissa; George Tzovaras, MD, Study Chair — University Hospital of Larissa; Georgia Stamatiou, MD, Study Director — University Hospital of Larissa; Elena Theodorou, MD, Study Chair — University Hospital of Larissa; Stavroula Georgopoulou, MD, Study Chair — University Hospital of Larissa
Locations (1):
- University Hospital of Larissa, Larissa, Greece

REFERENCES:
- [Background] Jokela R, Ahonen J, Tallgren M, Haanpaa M, Korttila K. A randomized controlled trial of perioperative administration of pregabalin for pain after laparoscopic hysterectomy. Pain. 2008 Jan;134(1-2):106-12. doi: 10.1016/j.pain.2007.04.002. Epub 2007 May 15. PMID 17507163
- [Background] White PF, Tufanogullari B, Taylor J, Klein K. The effect of pregabalin on preoperative anxiety and sedation levels: a dose-ranging study. Anesth Analg. 2009 Apr;108(4):1140-5. doi: 10.1213/ane.0b013e31818d40ce. PMID 19299776
- [Background] Paech MJ, Goy R, Chua S, Scott K, Christmas T, Doherty DA. A randomized, placebo-controlled trial of preoperative oral pregabalin for postoperative pain relief after minor gynecological surgery. Anesth Analg. 2007 Nov;105(5):1449-53, table of contents. doi: 10.1213/01.ane.0000286227.13306.d7. PMID 17959981
- [Background] Mathiesen O, Rasmussen ML, Dierking G, Lech K, Hilsted KL, Fomsgaard JS, Lose G, Dahl JB. Pregabalin and dexamethasone in combination with paracetamol for postoperative pain control after abdominal hysterectomy. A randomized clinical trial. Acta Anaesthesiol Scand. 2009 Feb;53(2):227-35. doi: 10.1111/j.1399-6576.2008.01821.x. Epub 2008 Dec 6. PMID 19076108
- [Background] Mathiesen O, Jacobsen LS, Holm HE, Randall S, Adamiec-Malmstroem L, Graungaard BK, Holst PE, Hilsted KL, Dahl JB. Pregabalin and dexamethasone for postoperative pain control: a randomized controlled study in hip arthroplasty. Br J Anaesth. 2008 Oct;101(4):535-41. doi: 10.1093/bja/aen215. Epub 2008 Jul 23. PMID 18653493
- [Background] Bisgaard T. Analgesic treatment after laparoscopic cholecystectomy: a critical assessment of the evidence. Anesthesiology. 2006 Apr;104(4):835-46. doi: 10.1097/00000542-200604000-00030. PMID 16571981
- [Background] Chang SH, Lee HW, Kim HK, Kim SH, Kim DK. An evaluation of perioperative pregabalin for prevention and attenuation of postoperative shoulder pain after laparoscopic cholecystectomy. Anesth Analg. 2009 Oct;109(4):1284-6. doi: 10.1213/ane.0b013e3181b4874d. Epub 2009 Jul 29. PMID 19641054
- [Background] Agarwal A, Gautam S, Gupta D, Agarwal S, Singh PK, Singh U. Evaluation of a single preoperative dose of pregabalin for attenuation of postoperative pain after laparoscopic cholecystectomy. Br J Anaesth. 2008 Nov;101(5):700-4. doi: 10.1093/bja/aen244. Epub 2008 Aug 20. PMID 18716003
- [Background] Cabrera Schulmeyer MC, de la Maza J, Ovalle C, Farias C, Vives I. Analgesic effects of a single preoperative dose of pregabalin after laparoscopic sleeve gastrectomy. Obes Surg. 2010 Dec;20(12):1678-81. doi: 10.1007/s11695-009-9944-1. Epub 2009 Aug 29. PMID 19727980
- [Background] Jokela R, Ahonen J, Tallgren M, Haanpaa M, Korttila K. Premedication with pregabalin 75 or 150 mg with ibuprofen to control pain after day-case gynaecological laparoscopic surgery. Br J Anaesth. 2008 Jun;100(6):834-40. doi: 10.1093/bja/aen098. Epub 2008 Apr 29. PMID 18448418
- [Background] Peng PW, Li C, Farcas E, Haley A, Wong W, Bender J, Chung F. Use of low-dose pregabalin in patients undergoing laparoscopic cholecystectomy. Br J Anaesth. 2010 Aug;105(2):155-61. doi: 10.1093/bja/aeq116. Epub 2010 Jun 25. PMID 20581215
- [Background] Ittichaikulthol W, Virankabutra T, Kunopart M, Khamhom W, Putarawuthichai P, Rungphet S. Effects of pregabalin on post operative morphine consumption and pain after abdominal hysterectomy with/without salphingo-oophorectomy: a randomized, double-blind trial. J Med Assoc Thai. 2009 Oct;92(10):1318-23. PMID 19845240
- [Background] Gajraj NM. Pregabalin: its pharmacology and use in pain management. Anesth Analg. 2007 Dec;105(6):1805-15. doi: 10.1213/01.ane.0000287643.13410.5e. PMID 18042886
- [Result] Sarakatsianou C, Theodorou E, Georgopoulou S, Stamatiou G, Tzovaras G. Effect of pre-emptive pregabalin on pain intensity and postoperative morphine consumption after laparoscopic cholecystectomy. Surg Endosc. 2013 Jul;27(7):2504-11. doi: 10.1007/s00464-012-2769-3. Epub 2013 Jan 24. PMID 23344509